CLINICAL TRIAL: NCT06309667
Title: A Double-blind, Randomized, Placebo Controlled, Combined Single (Part A) and Multiple (Part B, C) Ascending Dose, Phase 1 Study to Investigate the Safety, Tolerability and Pharmacokinetic and Pharmacodynamics Following Subcutaneous Injections of PG-102(MG12) in Healthy Adult and Obesity Participants
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics and Pharmacodynamics Following Subcutaneous Injections of PG-102 (MG12) in Healthy Adult and Obesity Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ProGen. Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SL-MG12-P1
Record Dates: First submitted 2024-02-14; First posted 2024-03-13 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (11):
- Cohort A1 - Single Ascending Dose (Experimental): PG-102(MG12) Dose 1 (N=8) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo
- Cohort A2 - Single Ascending Dose (Experimental): PG-102(MG12) Dose 2 (N=8) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo
- Cohort A3 - Single Ascending Dose (Experimental): PG-102(MG12) Dose 3 (N=8) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo
- Cohort A4 - Single Ascending Dose (Experimental): PG-102(MG12) Dose 4 (N=8) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo
- Cohort A5 - Multiple Ascending Dose (Experimental): PG-102(MG12) Dose 5 (N=8) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo
- Cohort B1 - Multiple Ascending Dose (Experimental): PG-102(MG12) Dose 1 (N=6) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo
- Cohort B2 - Multiple Ascending Dose (Experimental): PG-102(MG12) Dose 1~5 (N=6) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo
- Cohort B3 - Multiple Ascending Dose (Experimental): PG-102(MG12) Dose 1~5 (N=6) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo
- Cohort S - Multiple Ascending Dose (Experimental): PG-102(MG12) Optimal Dose (N=6) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo
- Cohort C1 - Multiple Ascending Dose (Experimental): PG-102(MG12) Dose 1 (N=12) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo
- Cohort C2 - Multiple Ascending Dose (Experimental): PG-102(MG12) Dose 1 (N=12) Subcutaneous injection
  Interventions: Drug: PG-102(MG12); Other: Placebo

INTERVENTIONS:
Drug: PG-102(MG12) — GLP-1 and GLP-2 fusion protein
Other: Placebo — Placebo drug of PG-102(MG12)

SUMMARY:
This is a Phase 1, first-in-human (FIH), randomized, double-blind, placebo-controlled, combined single (Part A) multiple (Part B, C) ascending dose, phase 1 study to investigate the safety, tolerability and pharmacokinetic and pharmacodynamics following subcutaneous injections of PG-102(MG12) in healthy adult participants.

This study will be conducted in 3 Parts (Part A, B and C), with up to 5 cohorts in each part.

DETAILED DESCRIPTION:
Part A (SAD):

In Part A, subjects will receive a single dose of study drug, and the safety and efficacy of PG-102(MG12) will be evaluated in healthy subjects.

Part B (MAD):

In Part B, subjects will receive once-weekly doses of the study drug for 4 weeks, and the safety and efficacy of PG-102(MG12) will be evaluated in otherwise healthy overweight adult subjects.

Part C (MAD):

In Part C, obese participants will receive five repeated subcutaneous doses of the study drug, and the safety and tolerability of PG-102 (MG12) will be assessed across two cohorts based on prior safety data from Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, aged 18 to 65 years inclusive at the time of signing informed consent
2. Body mass index (BMI) of 18 to 30kg/m2 (inclusive) for Part A, Body mass index (BMI) of 25 to 30kg/m2 (inclusive) for Part B and Body mass index (BMI) 30 kg/m² or higher for Part C

[Exclusion Criteria]

1. History of administration of prescription drugs, herbal medicines, over-the-counter drugs, or vitamin supplements within 10 days prior to the study or history of the following drugs and/or other foods within 90 days prior to screening:

   * Drugs that affect body weight (such as obesity medications, psychiatric drugs, beta blockers, diuretics, contraceptives, female hormones, proton-pump inhibitors (PPIs), H2 receptor antagonists, health functional foods/supplements, and formulas designed for weight control).
   * Drugs that have the potential to impact blood sugar, liver fat, and intestinal microorganisms (including GLP-1 receptor agonists, DPP-4 inhibitors, SGLT-2 inhibitors, thiazolidinediones (TZDs), fish oil, polyunsaturated fatty acids (PUFA), and ursodeoxycholic acid (UDCA)), as well as individuals who are currently using insulin.
2. History of gastrointestinal diseases (Crohn's disease, ulcers, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (excluding simple appendectomy or hernia surgery) that may affect the absorption of clinical trial drugs.
3. History of acute proliferative retinopathy or maculopathy, severe gastroparesis, and/or severe neuropathy.
4. History of surgical treatment for obesity within 2 years (example: bariatric surgery, gastric banding etc) or gastrointestinal procedures for weight loss (including LAP-BAND®), or uncontrolled gastrointestinal disorders at Screening (e.g., peptic ulcer, gastroesophageal reflux disease).

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) for Part A | Baseline to Day 29
  Number of participants with treatment-emergent adverse events (TEAEs)
Number of participants with treatment-emergent adverse events (TEAEs) for Part B | Baseline to Day 57
  Number of participants with treatment-emergent adverse events (TEAEs)
Number of participants with Serious adverse events (SAEs) as assessed by CTCAE v5.0 for Part A | Baseline to Day 29
  Number of participants with Serious adverse events (SAEs) as assessed by CTCAE v5.0
Number of participants with Serious adverse events (SAEs) as assessed by CTCAE v5.0 for Part B | Baseline to Day 57
  Number of participants with Serious adverse events (SAEs) as assessed by CTCAE v5.0
Number of participants with clinically significant abnormalities in vital signs for Part A | Baseline to Day 29
  Blood pressure (mmHg), Respiration (breathing) rate per minute, Body temperature (Celsius)
Number of participants with clinically significant abnormalities in vital signs for Part B | Baseline to Day 57
  Blood pressure (mmHg), Respiration (breathing) rate per minute, Body temperature (Celsius)
Number of participants with clinically significant abnormalities in 12-lead ECGs for Part A | Baseline to Day 29
  Ventricular rate (bpm), PR interval (msec), QRSD (msec), QT (msec), QTc (msec)
Number of participants with clinically significant abnormalities in 12-lead ECGs for Part B | Baseline to Day 57
  Ventricular rate (bpm), PR interval (msec), QRSD (msec), QT (msec), QTc (msec)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) for Part A | Baseline to Day 29
  Maximum plasma concentration (Cmax)
Maximum plasma concentration (Cmax) for Part B | Baseline to Day 57
  Maximum plasma concentration (Cmax)
Time to maximum plasma concentration (tmax) for Part A | Baseline to Day 29
  Time to maximum plasma concentration (tmax)
Time to maximum plasma concentration (tmax) for Part B | Baseline to Day 57
  Time to maximum plasma concentration (tmax)
Area under the concentration-time curve up to the last quantifiable time-point (AUC0-t) for Part A | Baseline to Day 29
  Area under the concentration-time curve up to the last quantifiable time-point (AUC0-t)
Area under the concentration-time curve up to the last quantifiable time-point (AUC0-t) for Part B | Baseline to Day 57
  Area under the concentration-time curve up to the last quantifiable time-point (AUC0-t)
Terminal half-life (t1/2) for Part A | Baseline to Day 29
  Terminal half-life (t1/2)
Terminal half-life (t1/2) for Part B | Baseline to Day 57
  Terminal half-life (t1/2)
Apparent total clearance (CL/F) for Part A | Baseline to Day 29
  Apparent total clearance (CL/F)
Apparent total clearance (CL/F) for Part B | Baseline to Day 57
  Apparent total clearance (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Seunghoon Han, MD, Principal Investigator — Catholic University Seoul St.Mary Hospital
Locations (1):
- Catholic University Seoul St.Mary Hospital,, Seocho, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No